CLINICAL TRIAL: NCT06426654
Title: Sintilimab Combined With Low-dose Radiation Therapy for Neoadjuvant Treatment of Locally Advanced Deficient Mismatch Repair/Microsatellite Instability-high Gastric Cancer: a Prospective, Multi-center, Single-arm, Phase Ib/II Clinical Trial
Brief Title: Sintilimab Combined With LDRT for Neoadjuvant Treatment of Locally Advanced dMMR/MSI-H Gastric Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ming Liu, Clinical Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCH242145
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; neoadjuvant therapy; sintilimab; LDRT
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sintilimab+LDRT (Experimental): Laparoscopic exploration is required in all patients to detect occult peritoneal metastases.
  All patients will start with one cycle of neoadjuvant therapy of sintilimab: 200 mg, iv drip, d1, q3w.
  Then, LDRT will be performed in the target area (including the primary gastric lesion and positive/suspected positive lymph nodes).
  After radiotherapy, patients will receive another three cycles of sintilimab. Radical D2 gastric cancer resection will be performed 4-6 weeks after the last administration of sintilimab.
  The adjuvant therapy will start in 4-6 weeks after the surgery, and we recommend adjuvant treatment with sintilimab for up to 10 cycles.
  Interventions: Drug: sintiliman plus LDRT

INTERVENTIONS:
Drug: sintiliman plus LDRT — All patients will start with one cycle of neoadjuvant therapy of sintilimab: sintilimab 200 mg, iv drip, d1, q3w.
  LDRT will be performed in the target area. After radiotherapy, patients will receive another three cycles of sintilimab.
  Radical D2 gastric cancer resection will be performed 4-6 weeks after the last administration of sintilimab.
  The adjuvant therapy will start in 4-6 weeks after the surgery, and we recommend adjuvant treatment with sintilimab for up to 10 cycles.

SUMMARY:
Recently, growing evidences have suggested that immunotherapy represents a promising treatment option for the neoadjuvant treatment of locally advanced mismatch repair-deficient (dMMR)/microsatellite instability-high (MSI-H) gastric cancer. In this study, we will explore the efficacy and safety of sintilimab and LDRT in the neoadjuvant treatment for locally advanced dMMR/MSI-H G/GEJ cancer.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm, phase Ib/II trial. In the phase Ib, 4 cases will be enrolled in each treatment group. In the phase II study, a total of 33 patients will be enrolled. Eligible patients will be registered and receive four cycles of sintilimab. Simultaneously, LDRT will be planned and administered. Radical D2 gastric cancer resection will be performed 4-6 weeks after the last administration of sintilimab. The primary endpoint of phase Ib is to determine the optimal radiation dose for phase II study. The primary endpoint of phase II is the pathological complete response (pCR) rate. Secondary endpoints include R0 resection rate, major pathological response (MPR), objective response rate (ORR), 3-year event-free survival (EFS) rate, 3-year overall survival (OS) rate and safety profile of the neoadjuvant regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years.
2. Histologically or cytologically confirmed diagnosis of locally advanced G/GEJ adenocarcinoma (cT2N+M0 or cT3-4aNanyM0) as assessed by exploratory laparoscopic surgery, ultrasonography and/or CT/MRI.
3. Resectable G/GEJ cancer, as judged by experienced surgeons.
4. dMMR and/or MSI-H.

4. Eastern Cooperative Oncology Group performance score (ECOG PS) ≤1. 5. Agree to provide blood, feces, and tissue specimens. 6. The expected survival is longer than 6 months. 7. There was no previous antitumor treatment (including chemotherapy, radiotherapy, targeted therapy, immunotherapy, interventional therapy, and other treatments with antitumor effects).

8. Adequate organ and hematological function. 9. Strict contraception. 10. Patients must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.

Exclusion Criteria:

1. Unable to comply with the research program or procedures.
2. Undergoing other drug clinical trials or having participated in any drug clinical trials one month before enrollment.
3. Active autoimmune disease or history of refractory autoimmune disease.
4. Receiving corticosteroids (> 10mg/d prednisone or equivalent dose of steroids) or other systematic immunosuppression therapies within 14 days before enrollment, excluding the following therapies: steroid hormone replacement therapy (≤10mg/d); local steroid therapy; and short-term, prophylactic steroid therapy for preventing allergies or nausea and vomiting.
5. Active or clinically significant cardiac disease:

   1. Congestive heart failure > New York Heart Association (NYHA) class 2;
   2. Active coronary artery disease;
   3. Arrhythmias requiring treatment other than β-blockers or digoxin;
   4. Unstable angina (with angina symptoms at rest), new angina within 3 months before enrollment, or new myocardial infarction within 6 months before enrollment
6. Other tumors that have not been treated or exist at the same time, except carcinoma in situ of the cervix, treated basal cell carcinoma or superficial bladder tumor. If the tumor was cured and no evidence of disease was found for more than 3 years, the patient can be enrolled. All other tumors must be treated at least 3 years before enrollment.
7. Patients with a history of HIV infection or active hepatitis B/C.
8. Ongoing > level 2 infection.
9. Symptomatic brain metastasis or meningioma.
10. Unhealed wounds, ulcers or fractures.
11. Renal failure patients requiring blood or peritoneal dialysis.
12. Epileptic that needs medication.
13. Active, symptomatic interstitial pneumonia, pleural or ascites that causes dyspnea (dyspnea ≥ 2 grade).
14. History of organ transplantation (including corneal transplantation).
15. Allergic to research drugs or similar drugs, or suspected allergies.
16. Pregnant or lactating women.
17. The investigator believes that patients who are not suitable for the study.
18. Medical, psychological or social conditions can affect the recruitment of patients and evaluation of study results.
19. Other antitumor therapy (chemotherapy, radiotherapy, surgery, immunotherapy, biotherapy, chemoembolization) other than investigator drugs. Palliative external irradiation for non-target lesions is allowed.
20. Previously used similar immune checkpoint inhibitors.
21. Major surgery 4 weeks before recruitment, open biopsy or major trauma surgery (excluding biliary stents, or percutaneous biliary drainage).
22. Treatment with antitumor Chinese herbal medicine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 5 months after the last subject participating in
  defined as the absence of viable tumor cells assessed by histological evaluation criteria after neoadjuvant therapy

SECONDARY OUTCOMES:
R0 resection rate | 5 months after the last subject participating in
  defined as the rate of the complete surgical removal of any residual cancer cells in the tumor bed
MPR rate | 5 months after the last subject participating in
  defined as tumor residual cells ≤10% in the surgical specimen
3-year event-free survival (DFS) | every 3 month postoperation up to 36 months
  defined as the proportion of patients without event 23 years after enrolment
2-year OS rate | every 3 month postoperation up to 36 months
  defined as the proportion of patients survived 3 years after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Kun Yang, M.D., Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: No